CLINICAL TRIAL: NCT00701233
Title: Evaluation of Intercarpal Botox Versus Steroid Injections for Carpal Tunnel Syndrome
Brief Title: Botulinum Toxin for Carpal Tunnel Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to generate MD's and patients for this study
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0708M13705
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Corticosteroid injection into Carpal Tunnel
  Interventions: Drug: Corticosteroid injection into Carpal Tunnel
- 1 (Active Comparator): Botulinum toxin injection into Carpal Tunnel
  Interventions: Drug: Botulinum toxin

INTERVENTIONS:
Drug: Botulinum toxin — 45 units Botox injected into Carpal Tunnel once
  Arms: 1
Drug: Corticosteroid injection into Carpal Tunnel — 40 mg Triamcinolone with one mL 1% lidocaine injected once into Carpal Tunnel
  Arms: 2

SUMMARY:
To compare local steroid injections to local Botulinum toxin A injection in a double-blinded study.

DETAILED DESCRIPTION:
To compare local steroid injections to local Botulinum toxin A injection in a double-blinded study. The goal is to investigate if Botulinum toxin A injections are effective for Carpal Tunnel Syndrome compared to steroid injections in terms of pain relief and length of symptom alleviation.

ELIGIBILITY:
Inclusion Criteria:

* Any individual with symptoms of carpal tunnel syndrome and a diagnosis of CTS either clinically or via EMG will be included into this study. There will be a total of 20 subjects displaying symptoms of CTS. The gender of the subjects will not determine enrollment. There is no requirement of male to female ratio for this study. There is no age cut-off or minimal age requirement to enroll in the study. No specific Racial or ethnic restrictions will be present for this study. Female subjects of childbearing potential (not surgically sterile or postmenopausal for at least 2 years) must have a negative pregnancy test at screening.

Exclusion Criteria:

1. Any individual who has a diagnosis of CTS (by EMG or other means) but no symptoms of CTS will be excluded from this study.
2. Vulnerable subjects as defined as children, pregnant women, those with limited autonomy, decisional incapacity and prisoners will not be enrolled in this study.
3. Individuals with any history of carpal tunnel release surgery and recurrent or persistent symptoms will be excluded form this study.
4. Subject is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | one week, one month, three months, six month, nine months, and twelve months

SECONDARY OUTCOMES:
Carpal Tunnel Syndrome Assessment Questionnaire | one week, one month, three months, six month, nine months, and twelve months

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Dykstra, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota PM&R Department, Minneapolis, Minnesota, United States